CLINICAL TRIAL: NCT01932957
Title: A RANDOMISED TRIAL COMPARING LAPARASCOPY VERSUS LAPAROTOMY IN THE MANAGEMENT OF WOMEN DIAGNOSED WITH ECTOPIC PREGNANCY
Brief Title: Laparascopy Versus Laparatomy in the Management of Ruptured Ectopic Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pretoria (Other)
Responsible Party: Principal Investigator, Leon Snyman, Professor, University of Pretoria
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ectopic Trial
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Ruptured Ectopic Pregnancy
Keywords: Laparoscopy; Ruptured ectopic pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparotomy arm (Other): Standard treatment
  Interventions: Procedure: Laparotomy arm
- Laparoscopy arm (Experimental): Treatment by laparoscopy
  Interventions: Procedure: Laparoscopy arm

INTERVENTIONS:
Procedure: Laparotomy arm — Laparotomy as standard treatment for ruptured ectopic pregnancy
  Arms: Laparotomy arm
Procedure: Laparoscopy arm — Laparoscopy as treatment for ruptured ectopic pregnancy
  Arms: Laparoscopy arm

SUMMARY:
Standard management for patients with ruptured ectopic pregnancies at our institution is treatment by laparotomy. This trail will investigate the feasibility of treatment with laparoscopy and will look at outcomes such as hospital stay and pain experienced

The hypothesis is that laparoscopy is a feasible treatment option associated with shorter hospital stay and less pain

DETAILED DESCRIPTION:
Laparoscopic surgery for the surgical management of women diagnosed with ectopic pregnancies has become the standard of care in many institutions around the world. Laparotomy is still the standard of care at Kalafong Hospital. There is very little high quality evidence with regard to the optimal surgical management approach for women with ruptured ectopic pregnancies.

The study aims to compare laparotomy with laparoscopy in this group of women with regards to outcomes such as length of hospital stay, number of days off work and pain.

This randomised study will be conducted at Kalafong hospital, on 140 patients diagnosed with ruptured ectopic pregnancy who are haemodynamically stable and are able and willing to provide informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Able to give informed consent
* must have two of the following three:
* systolic blood pressure >90 mmHg
* pulse rate <100 beats per minute
* heamoglobin >8 g/dL

Exclusion Criteria:

* <18 years
* haemodynamically unstable
* not able to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-05-02 (Actual); Primary Completion 2013-10-31 (Actual); Study Completion 2013-11-30 (Actual)

PRIMARY OUTCOMES:
Hospital stay | 5 days
  Hospital stay will be compared between the two groups

SECONDARY OUTCOMES:
Pain scores | 24 hours
  Pain scores b means of visual analog pain scale
Theatre time | 1 day
  Theatre times will be measured and compared for the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Leon C Snyman, MBChB FCOG, Principal Investigator — Principal Specialist, Department Obstetrics & Gynaecology, University of Pretoria
Locations (1):
- Kalafong Academic Hospital, Pretoria, Gauteng, South Africa